CLINICAL TRIAL: NCT07013877
Title: Evaluation of the Impact of the Use of RELAX Glasses on Patients' Anxiety During Invasive Care in Intensive Care, Post-operative Intensive Care and Continuous Monitoring
Brief Title: Audiovisual Distraction in Intensive Care
Acronym: DARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-02-03
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anxiety
Keywords: Audiovisual sedation; anxiety; resuscitation; post-operative intensive care; invasive care; continuous monitoring
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Group with RELAX glasses" (Experimental): To facilitate immersion, RELAX goggles will be placed on the patient if he or she has been randomized to the "RELAX Goggles Group" immediately after the investigator's assessment of anxiety and pain.
  During the use of RELAX glasses, content will be proposed:
  * Regional reports. The choice of region will be left to the patient.
  * Animal reports. The choice will be left to the patient.
  * Relaxation videos. The choice will be left to the patient.
  RELAX glasses will be removed at the end of the invasive treatment.
  Interventions: Behavioral: RELAX glasses
- Control group without glasses RELAX (No Intervention): Nothing more happens than the usual treatment

INTERVENTIONS:
Behavioral: RELAX glasses — Glasses which are a solution of audiovisual sedation by positiv distraction for hospital medical use
  Arms: "Group with RELAX glasses"

SUMMARY:
Resuscitation patients are subject to constant stress of multifactorial origin: their state of health, the noisy environment of critical care, the multiple examinations and care provided, lack of sleep, stress from their loved ones... It is estimated that 60% of resuscitation patients have experienced stress and 40% have been anxious during their hospitalization in intensive care. This permanent anxiety is punctuated by stress peaks, particularly at the time of invasive procedures frequently performed in the ICU.

This stress is said to have a negative impact on patients' ability to recover and on their length of stay in the ICU. What's more, these anxious symptoms can persist after hospitalization, leading to post-traumatic stress disorder. It therefore seems appropriate to find solutions aimed at reducing this stress.

Medication is often used to reduce stress and anxiety. Although effective, these molecules have undesirable side-effects and can also hinder the patient's recovery.

Alternative methods are already being studied as replacement or supplementary therapies to drugs. These include music therapy, aromatherapy, hypnosis and virtual reality.

Virtual reality has been used on resuscitation patients to improve tolerance to mechanical ventilation and to the resuscitation environment in general.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in intensive care, post-operative intensive care and continuous monitoring;
* Patient receiving invasive care placement of peripheral venous line, nasogastric tube insertion, bladder catheterization, dressing stage IV pressure sores, heavy dressing lasting > 15 minutes arterial gasometry by puncture;
* Patient of legal age;
* Patient with written consent;
* Patient with Glasgow score equal to 15;
* Socially insured patient;
* Patient willing to comply with all study procedures and duration.

Exclusion Criteria:

* Medical history contraindicating RELAX eyewear;
* Known and current abuse of alcohol and/or illicit drugs that may interfere with patient safety and/or compliance;
* Any condition that would make the patient unsuitable for the study: current presence of cognitive disorders (MMS < 15), severe psychiatric disorders (bipolar disorders, psychotic disorders according to DSM-V classification);
* Major anxiety requiring anxiolytic medication prior to invasive care;
* Patient under court protection;
* Patient participating in another study;
* Patient who has already participated in the DARE study.
* Patient's refusal to use glasses;
* Visually impaired or blind patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Show that the use of RELAX glasses reduces anxiety in patients undergoing invasive care in the intensive care unit, postoperative intensive care unit and continuous care unit (experimental group), compared with patients undergoing usual care without R | Patient anxiety will be assessed by the investigator immediately after the treatment has been explained. As soon as the invasive treatment has been completed, regardless of the randomization group, the investigator will reassess the patient's anxiety
  The difference in anxiety between the 2 groups will be measured using a visual analog anxiety scale (A mark of 0 indicates 'no anxiety', a mark of 10 indicates 'maximum anxiety)

SECONDARY OUTCOMES:
To compare the evolution of patient pain during invasive care in intensive care, post-operative intensive care and continuous monitoring between the experimental group and the control group | Patient's pain will be assessed by the investigator immediately after the treatment has been explained. As soon as the invasive treatment has been completed, regardless of the randomization group, the investigator will reassess the patient's pain
  Change in pain level will be measured by the difference between before and after invasive care. Pain level will be measured using a visual analog scale (The score 0 expresses 'no pain', the score 10 reflects 'maximum imaginable pain)
To compare the number of placement attempts during invasive care in the ICU, post-operative intensive care and continuous monitoring, between the 2 groups | As soon as the invasive procedure has been completed, regardless of the randomization group, the investigator will also complete the document recording the number of trial(s) required to perform the invasive procedure
  Number of placement attempts during invasive care
Compare overall patient satisfaction after invasive care between experimental and control groups | Patient satisfaction will be asked immediately after the invasive treatment. An envelope will be given to the patient, who will be able to rate his or her overall satisfaction on a visual analog scale, without feeling influenced by the nurse
  Overall patient satisfaction will be measured by a visual analog scale (A score of 0 indicates 'not satisfied', while a score of 10 reflects 'maximum satisfaction)
To evaluate nursing staff satisfaction after invasive care in a patient wearing glasses | As soon as the invasive treatment has been completed, the nurse completes the satisfaction questionnary
  Nurse satisfaction will be assessed by a self-assessment questionnaire after each invasive procedure (A score of 0 means that it was 'not at all difficult', while a score of 10 means that it was 'extremely difficult)
Evaluate the impact of patient agitation on the performance of invasive care between the 2 groups | As soon as the invasive treatment has been completed, regardless of the randomization group, the investigator also completes the patient agitation evaluation questionnary.
  In the 2 groups, patient agitation during invasive care will be assessed using a questionnaire completed by the nursing staff
  1. The patient has not been agitated
  2. The patient was agitated but this had no impact on invasive care
  3. Patient agitation was the cause of a change in invasive care
  4. Patient agitation was the cause of a temporary suspension of invasive care
  5. The patient's agitation is too great to consider continuing the treatment.